CLINICAL TRIAL: NCT02305563
Title: A Phase 1/2, Open-label Randomized Study of Ulocuplumab (BMS-936564) in Combination With Low Dose Cytarabine in Subjects With Newly Diagnosed Acute Myeloid Leukemia
Brief Title: An Investigational Immuno-therapy Study of Ulocuplumab in Combination With Low Dose Cytarabine in Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business objectives have changed, slow accrual, the standard of care for the patient population changed and we were unable to accrue any longer.
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA212-016
Record Dates: First submitted 2014-11-27; First posted 2014-12-02 (Estimated); Results first posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia | interventions — ulocuplumab; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Ulocuplumab + low dose Cytarabine (Experimental): Ulocuplumab + low dose Cytarabine (LDAC) Phase 1 (escalation cohort) - closed for enrollment
  Interventions: Drug: BMS-936564; Drug: Cytarabine
- Ulocuplumab Dose A + low dose Cytarabine (Experimental): Ulocuplumab Dose A + low dose Cytarabine Phase 2 (expansion cohort)
  Interventions: Drug: BMS-936564; Drug: Cytarabine
- Ulocuplumab Dose B + low dose Cytarabine (Experimental): Ulocuplumab Dose B + low dose Cytarabine Phase 2 (expansion cohort)
  Interventions: Drug: BMS-936564; Drug: Cytarabine
- low dose Cytarabine only (Other): Low Dose Cytarabine only Phase 2 (expansion cohort)
  Interventions: Drug: BMS-936564; Drug: Cytarabine

INTERVENTIONS:
Drug: BMS-936564
  Other Names: Ulocuplumab; MDX-1338
Drug: Cytarabine

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of ulocuplumab in combination with low dose cytarabine in the treatment of Newly Diagnosed Acute Myeloid Leukemia (AML).

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Newly Diagnosed Acute Myeloid Leukemia (AML)
* Considered inappropriate for intensive remission induction therapy by an investigator
* Not eligible for stem cell transplantation

Exclusion Criteria:

* Acute promyelocytic leukemia
* Current Myelodysplastic syndrome only subjects
* Unstable angina or uncontrolled congestive heart failure
* Any other malignancy, excluding basal or squamous cell carcinoma of the skin, in situ melanoma, cervical carcinoma in situ, localized prostate cancer, or superficial bladder cancer stage 0, from which the subject has not been disease-free for at least 3 years
* Respiratory disease requiring continuous supplemental oxygen

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-01-27 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (35):
- United States (9):
  - Ucla Center Health Sci, Los Angeles, California
  - UF Health Cancer Center at Orlando Health, Orlando, Florida
  - Norton Cancer Institute, Louisville, Kentucky
  - NYU Langone Medical Center, New York, New York
  - Duke University Adult Bone Marrow Transplant Clinic, Durham, North Carolina
  - University Of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - The University Of Texas MD Anderson Cancer Center, Houston, Texas
  - Froedtert Hospital & Medical College of Wisconsin, Milwaukee, Wisconsin
- Brazil (5):
  - Liga Paranaense De Combate Ao Cancer Erasto Gaertner, Curitiba, Paraná
  - Instituto Do Cancer Mae De Deus / Cor Hospital Mae De Deus, Porto Alegre, Rio Grande do Sul
  - Fundacao Pio Xii Hosp Cancer De Barretos, Barretos, São Paulo
  - IEP Sao Lucas, São Paulo
  - Local Institution, São Paulo
- Local Institution, Halifax, Nova Scotia, Canada
- Local Institution, Hong Kong, China
- Israel (2):
  - Local Institution, Jerusalem
  - Local Institution, Tel Aviv
- Italy (4):
  - Azienda Ospedaliero Universitaria Policlinico Vittorio Emanuele, Catania
  - Local Institution, Milan
  - Azienda Ospedaliera Di Rilievo Nazionale A. Cardarelli, Napoli
  - Local Institution, Roma
- Japan (8):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Fukuyama-shi, Hiroshima
  - Local Institution, Isehara, Kanagawa
  - Local Institution, Hirakata-shi, Osaka
  - Local Institution, Bunkyo-ku, Tokyo
  - Local Institution, Shinagawa-ku, Tokyo
  - Local Institution, Shinjuku-Ku, Tokyo
  - Local Institution, Tachikawa, Tokyo
- Local Institution, Bucharest, Romania
- Local Institution, Seoul, South Korea
- Taiwan (3):
  - Local Institution, Kaohsiung City
  - Local Institution, New Taipei City
  - Local Institution, Taoyuan

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 6 participants in Phase 1 and 64 participants in Phase 2 (70 in total) were assigned to treatment. 2 participants randomized to the LDAC-only arm in Phase 2 did not receive treatment. 68 participants in total (phases 1 and 2) were treated.
Groups:
- ULO 600mg + LDAC - Ph1: Ulocuplumab (ULO) at 600mg + low dose cytarabine (LDAC) - Phase 1 (Ph1)
- ULO 800mg + LDAC - Ph1: Ulocuplumab (ULO) at 800mg + low dose cytarabine (LDAC) - Phase 1 (Ph1)
- ULO 800mg + LDAC - Ph2: Ulocuplumab (ULO) at 800mg + low dose cytarabine (LDAC) - Phase 2 (Ph2)
- ULO 1000mg + LDAC - Ph2: Ulocuplumab (ULO) at 1000mg + low dose cytarabine (LDAC) - Phase 2 (Ph2)
- LDAC - Ph2: Low dose cytarabine (LDAC) - Phase 2 (Ph2) Participants in the LDAC only arm were permitted to add ulocuplumab 800 mg into their treatment regimen if they did not achieve complete remission (CR or complete remission with incomplete blood count recovery [CRi]) confirmed by blast count reduction after 4 treatment cycles or if they relapsed after achieving complete remission
Period: Treatment Period
Arm/Group | ULO 600mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph2 | ULO 1000mg + LDAC - Ph2 | LDAC - Ph2
Started (Started = Randomized) | 3 | 3 | 26 | 14 | 24
Completed (Completed = Continuing in the treatment period) | 1 (At the time of the Phase 1 lock, 1 participant was still continuing on treatment) | 1 (At the time of the Phase 1 lock, 1 participant was still continuing on treatment) | 0 | 0 | 0
Not Completed | 2 | 2 | 26 | 14 | 24
Not completed — Disease progression | 0 | 0 | 15 | 6 | 6
Not completed — Study drug toxicity | 0 | 0 | 0 | 1 | 2
Not completed — Death | 0 | 0 | 1 | 2 | 1
Not completed — Adverse Event (AE) unrelated to drug | 0 | 0 | 7 | 1 | 2
Not completed — Participant request to stop therapy | 0 | 2 | 0 | 1 | 0
Not completed — Participant withdrew consent | 0 | 0 | 1 | 1 | 1
Not completed — Maximum clinical benefit | 0 | 0 | 0 | 0 | 1
Not completed — Poor/non-compliance | 0 | 0 | 0 | 0 | 1
Not completed — Administrative reason by Sponsor | 0 | 0 | 0 | 0 | 1
Not completed — other reason | 2 | 0 | 2 | 2 | 1
Not completed — Randomized but not treated | 0 | 0 | 0 | 0 | 2
Not completed — added ULO, then disease progression | 0 | 0 | 0 | 0 | 4
Not completed — added ULO; then other reason | 0 | 0 | 0 | 0 | 1
Not completed — added ULO, then request to stop | 0 | 0 | 0 | 0 | 1
Period: Follow-up Period
Arm/Group | ULO 600mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph2 | ULO 1000mg + LDAC - Ph2 | LDAC - Ph2
Started (Started = Entered follow-up) | 3 | 3 | 11 | 6 | 12
Completed (Completed = Continuing in the follow-up period) | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 11 | 6 | 12
Not completed — Death | 0 | 0 | 5 | 4 | 7
Not completed — Participant withdrew consent | 0 | 0 | 2 | 1 | 0
Not completed — other reason | 0 | 0 | 0 | 0 | 1
Not completed — Followup no longer required per protocol | 3 | 3 | 4 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ULO 600mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph2 | ULO 1000mg + LDAC - Ph2 | LDAC - Ph2 | Total
Number analyzed (Participants) | 3 | 3 | 26 | 14 | 24 | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.7 (8.02) | 77.3 (1.53) | 74.9 (5.4) | 73.1 (3.7) | 75.9 (5.7) | 74.9 (5.21)
Age, Customized [Number; unit: Participants] — Age categorical
  Participants
    <70 | 1 | 0 | 4 | 3 | 3 | 11
    >=70 | 2 | 3 | 22 | 11 | 21 | 59
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 9 | 7 | 14 | 33
  Male | 0 | 3 | 17 | 7 | 10 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: data not collected
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    White | 0 | 0 | 15 | 4 | 12 | 31
    Black/African American | 0 | 0 | 0 | 0 | 0 | 0
    Japanese | 3 | 3 | 6 | 6 | 4 | 22
    Chinese | 0 | 0 | 2 | 2 | 3 | 7
    Asian Indian | 0 | 0 | 0 | 0 | 0 | 0
    Asian Other | 0 | 0 | 3 | 0 | 2 | 5
    American Indian/Alaskan Native | 0 | 0 | 0 | 1 | 0 | 1
    Native Hawaiian/Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    Other | 0 | 0 | 0 | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs) in Treatment Cycle 1 - Phase 1
Description: Safety data evaluated for DLTs. DLTs and all other toxicities were defined and evaluated using the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.03 (NCI CTCAE v4.03). DLTs were defined based upon events that were considered to be related to ulocuplumab in combination with LDAC and that occurred during the first cycle of drug administration (28 days).
Time Frame: From first dose to end of cycle 1 (28 days)
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | ULO 600mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph1
Number analyzed (Participants) | 3 | 3
Participants | 0 | 0

2. Primary Outcome: Number of Participants With Adverse Events (AEs) - Phase 1
Description: The number of participants with an on-study adverse event (AE).
  Safety data are evaluated for AEs, defined and evaluated using the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.03 (NCI CTCAE v4.03).
Time Frame: From first dose to 30 days post last dose
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | ULO 600mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph1
Number analyzed (Participants) | 3 | 3
Participants | 3 | 3

3. Primary Outcome: Number of Participants With >= Grade 3 AEs - Phase 1
Description: The number of participants with an on-study adverse event >= Grade level 3.
  Safety data are evaluated for >= Grade 3 AEs, defined and evaluated using the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.03 (NCI CTCAE v4.03).
Time Frame: From first dose to 30 days post last dose
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | ULO 600mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph1
Number analyzed (Participants) | 3 | 3
Participants | 3 | 3

4. Primary Outcome: Number of Participants With AEs Leading to Discontinuation - Phase 1
Description: The number of participants with an on-study adverse event (AE) leading to discontinuation.
  Safety data are evaluated for AEs leading to discontinuation, defined and evaluated using the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.03 (NCI CTCAE v4.03).
Time Frame: From first dose to 30 days post last dose
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | ULO 600mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph1
Number analyzed (Participants) | 3 | 3
Participants | 0 | 0

5. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) - Phase 1
Description: The number of participants with an on-study serious adverse event (SAE).
  Safety data are evaluated for SAEs, defined and evaluated using the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.03 (NCI CTCAE v4.03).
Time Frame: From first dose to 30 days post last dose
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | ULO 600mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph1
Number analyzed (Participants) | 3 | 3
Participants | 2 | 1

6. Primary Outcome: Number of Deaths - Phase 1
Description: The number of participants who died.
Time Frame: From first dose to 30 days post last dose
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | ULO 600mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph1
Number analyzed (Participants) | 3 | 3
Participants | 0 | 0

7. Primary Outcome: Number of Participants With Laboratory Abnormalities - Phase 1
Description: The number of participants with an on-study laboratory abnormality.
  Safety data are evaluated for laboratory abnormalities, defined and evaluated using the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.03 (NCI CTCAE v4.03).
  grades 1, 2, 3, 4, 5, unknown, with 5 being the worst outcome
Time Frame: From first dose to 30 days post last dose
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | ULO 600mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph1
Number analyzed (Participants) | 3 | 3
Participants
  ABSOLUTE NEUTROPHIL COUNT - grade 3 | 0 | 1
  ABSOLUTE NEUTROPHIL COUNT - grade 4 | 3 | 2
  ALANINE AMINOTRANSFERASE - grade 0 | 2 | 2
  ALANINE AMINOTRANSFERASE - grade 1 | 1 | 1
  ALBUMIN - grade 0 | 1 | 0
  ALBUMIN - grade 1 | 0 | 2
  ALBUMIN - grade 2 | 2 | 1
  ALKALINE PHOSPHATASE - grade 0 | 2 | 2
  ALKALINE PHOSPHATASE grade 1 | 1 | 1
  ASPARTATE AMINOTRANSFERASE - grade 0 | 3 | 2
  ASPARTATE AMINOTRANSFERASE - grade 1 | 0 | 1
  BILIRUBIN, TOTAL - grade 0 | 3 | 2
  BILIRUBIN, TOTAL - grade 2 | 0 | 1
  CALCIUM, TOTAL - grade 0 | 1 | 1
  CALCIUM, TOTAL - grade 1 | 0 | 1
  CALCIUM, TOTAL - grade 2 | 2 | 1
  CREATINE KINASE - grade 0 | 3 | 3
  CREATININE - grade 0 | 2 | 3
  CREATININE - grade 1 | 1 | 0
  FIBRINOGEN - grade 0 | 1 | 0
  GLUCOSE, FASTING SERUM - grade 0 | 1 | 1
  GLUCOSE, FASTING SERUM - grade 1 | 2 | 0
  GLUCOSE, FASTING SERUM - grade 2 | 0 | 2
  HEMOGLOBIN - grade 2 | 1 | 1
  HEMOGLOBIN - grade 3 | 2 | 2
  LEUKOCYTES - grade 0 | 0 | 1
  LEUKOCYTES - grade 3 | 1 | 1
  LEUKOCYTES - grade 4 | 2 | 1
  LIPASE, TOTAL (COLORIMETRIC ASSAY) - grade 0 | 2 | 1
  LIPASE, TOTAL (COLORIMETRIC ASSAY) - grade 1 | 1 | 0
  LIPASE, TOTAL (COLORIMETRIC ASSAY) - grade 3 | 0 | 2
  LYMPHOCYTES (ABSOLUTE) - grade 0 | 0 | 1
  LYMPHOCYTES (ABSOLUTE) - grade 1 | 0 | 1
  LYMPHOCYTES (ABSOLUTE) - grade 2 | 2 | 1
  LYMPHOCYTES (ABSOLUTE) - grade 3 | 1 | 0
  NEUTROPHILS (ABSOLUTE) - grade 3 | 0 | 1
  NEUTROPHILS (ABSOLUTE) - grade 4 | 3 | 2
  PHOSPHORUS, INORGANIC - grade 0 | 3 | 2
  PHOSPHORUS, INORGANIC - grade 3 | 0 | 1
  PLATELET COUNT - grade 3 | 0 | 1
  PLATELET COUNT - grade 4 | 3 | 2
  POTASSIUM, SERUM - grade 0 | 1 | 2
  POTASSIUM, SERUM - grade 1 | 0 | 1
  POTASSIUM, SERUM - grade 3 | 2 | 0
  SODIUM, SERUM - grade 0 | 2 | 1
  SODIUM, SERUM - grade 1 | 0 | 2
  SODIUM, SERUM - grade 3 | 1 | 0
  URIC ACID - grade 0 | 3 | 2
  URIC ACID - grade 1 | 0 | 1

8. Primary Outcome: Best Overall Response (BOR) - Phase 2
Description: The phase 2 primary endpoint was based on the rate of Complete Remission (CR/CRi) prior to the initiation of any alternative therapy (including any subsequent ulocuplumab 800 mg for participants in the LDAC alone arm). The phase 2 primary analysis was conducted after all participants had an opportunity for 6 months of follow-up.
  Complete remission rate: CR + CRi, confidence interval based on the Clopper and Pearson method.
  CR = complete response CRi = complete response, incomplete blood count
Time Frame: From first dose until a minimum follow-up of up to 2 months
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ULO 800mg + LDAC - Ph2 | ULO 1000mg + LDAC - Ph2 | LDAC - Ph2
Number analyzed (Participants) | 26 | 14 | 24
Percentage of participants | 15.4 [4.4 to 34.9] | 7.1 [0.2 to 33.9] | 25.0 [9.8 to 46.7]

9. Secondary Outcome: Best Overall Response (BOR) - Phase 1
Description: Investigator assessed best overall response prior to the initiation of any alternative therapy for Phase 1 participants.
Time Frame: From first dose until a minimum follow-up of up to 2 months
Population: All randomized participants
Measure: Number; unit: Participants
Arm/Group | ULO 600mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph1
Number analyzed (Participants) | 3 | 3
Participants | 1 | 3

10. Secondary Outcome: Number of Participants With AEs - Phase 2
Description: as for outcome 2
Time Frame: From first dose until a minimum follow-up of up to 2 months
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | ULO 800mg + LDAC - Ph2 | ULO 1000mg + LDAC - Ph2 | LDAC - Ph2
Number analyzed (Participants) | 26 | 14 | 22
Participants | 25 | 14 | 22

11. Secondary Outcome: Number of Participants With AEs Leading to Discontinuation - Phase 2
Description: as for outcome 4
Time Frame: From first dose until a minimum follow-up of up to 2 months
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | ULO 800mg + LDAC - Ph2 | ULO 1000mg + LDAC - Ph2 | LDAC - Ph2
Number analyzed (Participants) | 26 | 14 | 22
Participants | 7 | 3 | 4

12. Secondary Outcome: Number of Participants With SAEs - Phase 2
Description: as for outcome 5
Time Frame: From first dose until a minimum follow-up of up to 2 months
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | ULO 800mg + LDAC - Ph2 | ULO 1000mg + LDAC - Ph2 | LDAC - Ph2
Number analyzed (Participants) | 26 | 14 | 22
Participants | 21 | 8 | 15

13. Secondary Outcome: Number of Deaths- Phase 2
Description: The number of participants who died.
  Safety data are evaluated for deaths, defined and evaluated using the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.03 (NCI CTCAE v4.03).
Time Frame: From first dose until a minimum follow-up of up to 2 months
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | ULO 800mg + LDAC - Ph2 | ULO 1000mg + LDAC - Ph2 | LDAC - Ph2
Number analyzed (Participants) | 26 | 14 | 22
Participants | 19 | 10 | 16

14. Secondary Outcome: Number of Participants With Laboratory Abnormalities - Phase 2
Description: The number of participants with an on-study laboratory abnormality, assessed from Grade 1-4 Serum Chemistry, Electrolytes, and Hematology Laboratory Test results, with grade 4 being the worst.
  Safety data are evaluated for laboratory abnormalities, defined and evaluated using the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.03 (NCI CTCAE v4.03).
Time Frame: From first dose until a minimum follow-up of up to 2 months
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | ULO 800mg + LDAC - Ph2 | ULO 1000mg + LDAC - Ph2 | LDAC - Ph2
Number analyzed (Participants) | 26 | 14 | 22
Participants
  ALANINE AMINOTRANSFERASE (ALT), grade 1 | 5 | 5 | 4
  ALANINE AMINOTRANSFERASE (ALT), grade 2 | 0 | 1 | 2
  ALANINE AMINOTRANSFERASE (ALT), grade 3 | 2 | 2 | 0
  ALKALINE PHOSPHATASE (ALP), grade 1 | 9 | 3 | 8
  ALKALINE PHOSPHATASE (ALP), grade 2 | 1 | 5 | 2
  ASPARTATE AMINOTRANSFERASE (AST), grade 1 | 7 | 8 | 4
  ASPARTATE AMINOTRANSFERASE (AST), grade 2 | 1 | 0 | 2
  ASPARTATE AMINOTRANSFERASE (AST), grade 3 | 0 | 1 | 0
  BILIRUBIN, TOTAL, grade 1 | 3 | 2 | 1
  BILIRUBIN, TOTAL, grade 2 | 4 | 3 | 1
  BILIRUBIN, TOTAL, grade 3 | 1 | 0 | 0
  CREATININE, grade 1 | 7 | 5 | 6
  CREATININE, grade 2 | 5 | 2 | 2
  CALCIUM, TOTAL, grade 1 | 7 | 3 | 3
  CALCIUM, TOTAL, grade 2 | 5 | 5 | 7
  CALCIUM, TOTAL, grade 3 | 0 | 1 | 0
  PHOSPHORUS, INORGANIC, grade 1 | 0 | 0 | 1
  PHOSPHORUS, INORGANIC, grade 2 | 3 | 2 | 1
  PHOSPHORUS, INORGANIC, grade 3 | 2 | 0 | 2
  PHOSPHORUS, INORGANIC, grade 4 | 0 | 1 | 0
  POTASSIUM, SERUM, grade 1 | 4 | 3 | 5
  POTASSIUM, SERUM, grade 2 | 0 | 1 | 0
  POTASSIUM, SERUM, grade 3 | 1 | 2 | 4
  POTASSIUM, SERUM, grade 4 | 1 | 1 | 0
  SODIUM, SERUM, grade 1 | 9 | 3 | 7
  SODIUM, SERUM, grade 2 | 0 | 1 | 0
  SODIUM, SERUM, grade 3 | 0 | 3 | 4
  HEMOGLOBIN, grade 2 | 2 | 4 | 4
  HEMOGLOBIN, grade 3 | 22 | 10 | 17
  PLATELET COUNT, grade 2 | 0 | 0 | 1
  PLATELET COUNT, grade 3 | 1 | 1 | 3
  PLATELET COUNT, grade 4 | 23 | 13 | 17
  ABSOLUTE NEUTROPHIL COUNT, grade 1 | 2 | 1 | 0
  ABSOLUTE NEUTROPHIL COUNT, grade 2 | 0 | 1 | 1
  ABSOLUTE NEUTROPHIL COUNT, grade 3 | 3 | 0 | 1
  ABSOLUTE NEUTROPHIL COUNT, grade 4 | 18 | 10 | 16
  LEUKOCYTES, grade 1 | 3 | 0 | 1
  LEUKOCYTES, grade 2 | 3 | 4 | 0
  LEUKOCYTES, grade 3 | 6 | 4 | 5
  LEUKOCYTES, grade 4 | 8 | 1 | 10
  LYMPHOCYTES (ABSOLUTE), grade 1 | 3 | 4 | 1
  LYMPHOCYTES (ABSOLUTE), grade 2 | 7 | 1 | 7
  LYMPHOCYTES (ABSOLUTE), grade 3 | 5 | 0 | 7
  LYMPHOCYTES (ABSOLUTE), grade 4 | 0 | 0 | 1
  NEUTROPHILS (ABSOLUTE), grade 1 | 1 | 0 | 0
  NEUTROPHILS (ABSOLUTE), grade 2 | 1 | 2 | 1
  NEUTROPHILS (ABSOLUTE), grade 3 | 3 | 0 | 1
  NEUTROPHILS (ABSOLUTE), grade 4 | 18 | 10 | 16

15. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA) Positive for Ulocuplumab - Phases 1 and 2
Description: Serum samples from ulocuplumab treated participants were evaluated for the presence of anti-ulocuplumab antibodies
Time Frame: From first dose until a minimum follow-up of up to 2 months
Population: All participants treated with ulocuplumab
Measure: Number; unit: Participants
Arm/Group | ULO 600mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph2 | ULO 1000mg + LDAC - Ph2
Number analyzed (Participants) | 3 | 3 | 21 | 14
Participants | 0 | 0 | 6 | 0

16. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) - Phases 1 and 2
Description: The Pharmacokinetic (PK) parameters are assessed for ulocuplumab following study drug administration
  EOT = end of treatment
  Measure type and method of dispersion are Geometric mean and %CV, respectively
Time Frame: Cycle 1 Day 1
Population: All treated participants who have evaluable PK profiles
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | ULO 600mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph2 | ULO 1000mg + LDAC - Ph2 | LDAC - Ph2
Number analyzed (Participants) | 3 | 3 | 17 | 14 | 1
µg/mL | 219.354 (19) | 265.294 (8) | 183.456 (25) | 256.906 (22) | 212.564 (NA) — Not applicable as n=1

17. Secondary Outcome: Trough Observed Serum Concentration (Ctrough) - Phases 1 and 2
Description: The Pharmacokinetic (PK) parameters are assessed for ulocuplumab following study drug administration.
  EOT = end of treatment
  Measure type and method of dispersion are Geometric mean and %CV, respectively
Time Frame: Days 1, 8, 15 for cycle 1; Days 8, 15 for cycle 2; Days 1, 8 for cycles 3-5; Day 1 every 4th cycle thereafter; EOT; 30 days post last dose (follow-up)
Population: All treated participants who have evaluable PK profiles
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | ULO 600mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph2 | ULO 1000mg + LDAC - Ph2 | LDAC - Ph2
Number analyzed (Participants) | 3 | 3 | 22 | 13 | 1
µg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 3 | 20 | 8 | 1
  Cycle 1 Day 1 | 0.100 (0) | 0.100 (0) | 0.100 (0) | 0.100 (0) | 0.100 (NA) — Not applicable as n=1
  Cycle 1 Day 8 | 5.308 (89) | 75.890 (30) | 10.321 (85) | 17.766 (79) | 39.609 (NA) — Not applicable as n=1
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 3 | 19 | 11 | 1
  Cycle 1 Day 15 | 21.748 (91) | 125.797 (18) | 37.263 (66) | 61.250 (64) | 175.315 (NA) — Not applicable as n=1
  Cycle 2 Day 8: number analyzed (Participants) | 1 | 3 | 15 | 10 | 0
  Cycle 2 Day 8 | 41.630 (NA) — Not applicable as n=1 | 96.333 (36) | 30.916 (83) | 103.322 (67) |
  Cycle 2 Day 15: number analyzed (Participants) | 1 | 3 | 14 | 8 | 0
  Cycle 2 Day 15 | 72.104 (NA) — Not applicable as n=1 | 126.029 (49) | 48.421 (73) | 143.724 (58) |
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 1 | 12 | 3 | 0
  Cycle 3 Day 1 |  | 78.218 (NA) — Not applicable as n=1 | 13.905 (101) | 153.871 (70) |
  Cycle 3 Day 8: number analyzed (Participants) | 1 | 3 | 11 | 3 | 0
  Cycle 3 Day 8 | 85.993 (NA) — Not applicable as n=1 | 129.580 (42) | 37.602 (94) | 82.033 (21) |
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 2 | 6 | 1 | 0
  Cycle 4 Day 1 |  | 80.409 (64) | 4.012 (145) | 212.793 (NA) — Not applicable as n=1 |
  Cycle 4 Day 8: number analyzed (Participants) | 1 | 3 | 3 | 2 | 0
  Cycle 4 Day 8 | 112.048 (NA) — Not applicable as n=1 | 133.650 (41) | 116.657 (83) | 77.095 (119) |
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 1 | 3 | 1 | 0
  Cycle 5 Day 1 |  | 32.621 (NA) — Not applicable as n=1 | 4.558 (166) | 224.703 (NA) — Not applicable as n=1 |
  Cycle 5 Day 8: number analyzed (Participants) | 1 | 2 | 3 | 1 | 0
  Cycle 5 Day 8 | 102.751 (NA) — Not applicable as n=1 | 124.996 (48) | 34.783 (137) | 202.552 (NA) — Not applicable as n=1 |
  Cycle 9 Day 1: number analyzed (Participants) | 0 | 0 | 2 | 1 | 0
  Cycle 9 Day 1 |  |  | 35.144 (110) | 187.930 (NA) — Not applicable as n=1 |
  EOT: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  EOT |  |  | 0.100 (NA) — Not applicable as n=1 |  |

18. Secondary Outcome: Time of Maximum Observed Ulocuplumab Serum Concentration (Tmax) - Phases 1 and 2
Description: The Pharmacokinetic (PK) parameters are assessed for ulocuplumab following study drug administration.
  EOT = end of treatment
Time Frame: Cycle 1 Day 1
Population: All treated participants who have evaluable PK profiles
Measure: Median (Full Range); unit: hour (H)
Arm/Group | ULO 600mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph2 | ULO 1000mg + LDAC - Ph2 | LDAC - Ph2
Number analyzed (Participants) | 3 | 3 | 17 | 7 | 1
hour (H) | 1.850 [1.47 to 2.02] | 1.933 [1.68 to 2.03] | 1.500 [1.00 to 4.50] | 2.117 [1.28 to 5.12] | 2.03 [2.03 to 2.03]

19. Secondary Outcome: Area Under the Ulocuplumab Concentration-time Curve From Time Zero to the Last Quantifiable Concentration [AUC(0-T)] - Phases 1 and 2
Description: The Pharmacokinetic (PK) parameters are assessed for ulocuplumab following study drug administration.
  EOT = end of treatment
  AUC(0-T) calculated by log- and linear-trapezoidal summation
  Measure type and method of dispersion are Geometric mean and %CV, respectively
Time Frame: Cycle 1 Day 1
Population: All treated participants who have evaluable PK profiles
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg.h/mL
Arm/Group | ULO 600mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph2 | ULO 1000mg + LDAC - Ph2 | LDAC - Ph2
Number analyzed (Participants) | 3 | 3 | 17 | 7 | 1
µg.h/mL | 9455.529 (10) | 21158.725 (9) | 8152.698 (50) | 13744.382 (37) | 16502.463 (NA) — Not applicable as n=1

20. Secondary Outcome: Area Under the Ulocuplumab Concentration-time Curve in One Dosing Interval [AUC(TAU)] - Phases 1 and 2
Description: as for outcome 17
Time Frame: Cycle 1 Day 1
Population: All treated participants who have evaluable PK profiles
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg.h/mL
Arm/Group | ULO 600mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph2 | ULO 1000mg + LDAC - Ph2 | LDAC - Ph2
Number analyzed (Participants) | 3 | 3 | 13 | 7 | 1
µg.h/mL | 9455.529 (10) | 21158.725 (9) | 10082.624 (38) | 13826.833 (36) | 14257.807 (NA) — Not applicable as n=1

21. Secondary Outcome: Area Under the Ulocuplumab Concentration-time Curve From Time Zero to Infinity [AUC(INF)] - Phases 1 and 2
Description: The Pharmacokinetic (PK) parameters are assessed for ulocuplumab following study drug administration.
  EOT = end of treatment
  AUC(INF) calculated by summing AUC(0-T) and the extrapolated area, computed by the quotient Clast/λz
  Measure type and method of dispersion are Geometric mean and %CV, respectively
Time Frame: Days 1, 8, 15 for cycles 1 and 2; Days 1, 8 for cycles 3-5; Day 1 every 4th cycle thereafter; EOT; 30 days post last dose (follow-up)
Population: Based on the PK sample collections, PK parameters depended on terminal phase time points including AUC(INF), T-HALF; or at steady-state, including CLT, Vss are not reportable
Arm/Group | ULO 600mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph2 | ULO 1000mg + LDAC - Ph2 | LDAC - Ph2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Elimination Half-life (T-HALF) - Phases 1 and 2
Description: The Pharmacokinetic (PK) parameters are assessed for ulocuplumab following study drug administration.
  EOT = end of treatment
  T-HALF determined as 0.693/λz
Time Frame: as for outcome 21
Population: as for outcome 21
Arm/Group | ULO 600mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph2 | ULO 1000mg + LDAC - Ph2 | LDAC - Ph2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Total Body Clearance of Ulocuplumab (CLT) - Phases 1 and 2
Description: The Pharmacokinetic (PK) parameters are assessed for ulocuplumab following study drug administration.
  EOT = end of treatment
  CLT calculated by dividing the total dose of ulocuplumab by its corresponding AUC(INF) value
  Measure type and method of dispersion are Geometric mean and %CV, respectively
Time Frame: as for outcome 21
Population: as for outcome 21
Arm/Group | ULO 600mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph2 | ULO 1000mg + LDAC - Ph2 | LDAC - Ph2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Volume of Distribution at Steady State (Vss) - Phases 1 and 2
Description: as for outcome 17
Time Frame: as for outcome 21
Population: as for outcome 21
Arm/Group | ULO 600mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph2 | ULO 1000mg + LDAC - Ph2 | LDAC - Ph2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Overall Rate of Remission in Participants Treated With Ulocuplumab at Two Different Dose Levels 800 mg and 1000 mg in Combination With LDAC - Phase 2
Description: This phase 2 secondary endpoint was based on the rate of Overall Remission (OR=PR+CR +CRi) prior to the initiation of any alternative therapy (including any subsequent ulocuplumab 800 mg for participants in the LDAC alone arm). The phase 2 analysis was conducted after all participants had an opportunity for 6 months of follow-up.
  Overall remission rate: CR + CRi, + PR confidence interval based on the Clopper and Pearson method.
  CR = complete response CRi = complete response, incomplete blood count PR = partial remission
Time Frame: From first dose until a minimum follow-up of up to 2 months
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ULO 800mg + LDAC - Ph2 | ULO 1000mg + LDAC - Ph2
Number analyzed (Participants) | 26 | 14
Percentage of participants | 19.2 [6.6 to 39.4] | 7.1 [0.2 to 33.9]

26. Secondary Outcome: Duration of Response in Participants With CR/CRi Treated With Ulocuplumab at Two Different Dose Levels 800 mg and 1000 mg in Combination With LDAC - Phase 2
Description: This phase 2 secondary endpoint was based on the duration of complete remission prior to the initiation of any alternative therapy (including any subsequent ulocuplumab 800 mg for participants in the LDAC alone arm). The phase 2 analysis was conducted after all participants had an opportunity for 6 months of follow-up.
Time Frame: From first dose until a minimum follow-up of up to 2 months
Population: All randomized participants with CR/CRi
Measure: Median (Full Range); unit: Months
Arm/Group | ULO 800mg + LDAC - Ph2 | ULO 1000mg + LDAC - Ph2
Number analyzed (Participants) | 4 | 1
Months | 2.4 [0.5 to 5.6] | 4.3 [NA to NA] — Only 1 participant

27. Secondary Outcome: Rate of Complete Remission (CR/CRi) and Overall Rate of Remission in Participants Treated With LDAC Only - Phase 2
Description: This phase 2 secondary endpoint was based on the rate of Complete Remission (CR/CRi) and rate of Overall Remission (OR=PR+CR +CRi) prior to the initiation of any alternative therapy (including any subsequent ulocuplumab 800 mg for participants in the LDAC alone arm). The phase 2 analysis was conducted after all participants had an opportunity for 6 months of follow-up.
  Overall remission rate: CR + CRi, + PR confidence interval based on the Clopper and Pearson method.
  CR = complete response CRi = complete response, incomplete blood count PR = partial remission
Time Frame: From first dose until a minimum follow-up of up to 2 months
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LDAC - Ph2
Number analyzed (Participants) | 24
Percentage of participants
  CR/CRi | 25.0 [9.8 to 46.7]
  Overall remission rate | 25.0 [9.8 to 46.7]

28. Secondary Outcome: Duration of Response in Participants With CR/CRi Treated With LDAC Only - Phase 2
Description: as for outcome 26
Time Frame: From first dose until a minimum follow-up of up to 2 months
Population: All randomized participants with CR/CRi
Measure: Median (Full Range); unit: Months
Arm/Group | LDAC - Ph2
Number analyzed (Participants) | 6
Months | 5.7 [0.9 to NA] — upper limit not reached

29. Secondary Outcome: Change From Baseline of Electrocardiogram (ECG) Endpoints: Heart Rate - Phases 1 and 2
Description: Change from baseline of ECG endpoints
  Heart rate measured in beats per minute (bpm)
Time Frame: From first dose until a minimum follow-up of up to 2 months
Population: All treated participants
Measure: Mean (Standard Deviation); unit: change from baseline bpm
Arm/Group | ULO 600mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph2 | ULO 1000mg + LDAC - Ph2 | LDAC - Ph2
Number analyzed (Participants) | 3 | 3 | 15 | 13 | 9
change from baseline bpm
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 2 | 15 | 13 | 9
  Cycle 2 Day 1 | 26.0 (63.6) | 4.0 (18.4) | 1.8 (11.3) | -0.9 (20.0) | -3.0 (7.6)
  Cycle 3, Day 1: number analyzed (Participants) | 3 | 2 | 13 | 6 | 7
  Cycle 3, Day 1 | -2.3 (18.8) | 0.0 (15.6) | 5.8 (14.2) | 12.7 (14.3) | 1.7 (10.2)
  Cycle 4, Day 1: number analyzed (Participants) | 1 | 2 | 9 | 3 | 7
  Cycle 4, Day 1 | -1.0 | -16.0 (5.7) | -0.1 (9.9) | 11.0 (40.6) | 1.3 (16.7)
  Cycle 5, Day 1: number analyzed (Participants) | 1 | 2 | 6 | 2 | 5
  Cycle 5, Day 1 | -6.0 | 1.5 (7.8) | 4.3 (12.3) | 10.5 (2.1) | 8.8 (27.5)
  Cycle 6, Day 1: number analyzed (Participants) | 1 | 3 | 4 | 0 | 7
  Cycle 6, Day 1 | -6.0 | -6.0 (16.5) | 6.8 (5.3) |  | 7.4 (14.9)
  Cycle 7, Day 1: number analyzed (Participants) | 0 | 3 | 4 | 1 | 6
  Cycle 7, Day 1 |  | -11.7 (18.6) | -3.5 (5.9) | 12.0 (NA) — Not applicable as n=1 | 6.5 (13.5)
  Cycle 8, Day 1: number analyzed (Participants) | 1 | 0 | 3 | 1 | 5
  Cycle 8, Day 1 | -1.0 |  | 0.7 (2.1) | 11.0 (NA) — Not applicable as n=1 | 0.8 (11.4)
  Cycle 9, Day 1: number analyzed (Participants) | 0 | 2 | 2 | 1 | 5
  Cycle 9, Day 1 |  | -17.0 (11.3) | 7.0 (7.1) | 3.0 (NA) — Not applicable as n=1 | 0.6 (8.9)
  Cycle 10, Day 1: number analyzed (Participants) | 1 | 1 | 3 | 0 | 2
  Cycle 10, Day 1 | -3.0 | -16.0 (NA) — Not applicable as n=1 | 9.3 (5.1) |  | 2.0 (1.4)
  Cycle 11, Day 1: number analyzed (Participants) | 1 | 0 | 0 | 1 | 3
  Cycle 11, Day 1 | -12.0 |  |  | 10.0 (NA) — Not applicable as n=1 | -0.3 (6.7)
  Cycle 12, Day 1: number analyzed (Participants) | 0 | 0 | 1 | 1 | 2
  Cycle 12, Day 1 |  |  | 5.0 (NA) — Not applicable as n=1 | 19.0 (NA) — Not applicable as n=1 | 7.0 (2.8)
  Cycle 13, Day 1: number analyzed (Participants) | 1 | 0 | 1 | 0 | 2
  Cycle 13, Day 1 | -9.0 |  | 8.0 (NA) — Not applicable as n=1 |  | 4.0 (2.8)
  Cycle 14, Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Cycle 14, Day 1 |  |  | 14.0 (NA) — Not applicable as n=1 |  |
  Cycle 15, Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1
  Cycle 15, Day 1 | -10.0 |  |  |  | 8.0 (NA) — Not applicable as n=1
  Cycle 16, Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Cycle 16, Day 1 |  |  |  |  | 18.0 (NA) — Not applicable as n=1

30. Secondary Outcome: Change From Baseline of Electrocardiogram (ECG) Endpoints: PR Interval - Phases 1 and 2
Description: Change from baseline of ECG endpoints
  PR interval measured in milliseconds (msec)
Time Frame: From first dose until a minimum follow-up of up to 2 months
Population: All treated participants
Measure: Mean (Standard Deviation); unit: change from baseline msec
Arm/Group | ULO 600mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph2 | ULO 1000mg + LDAC - Ph2 | LDAC - Ph2
Number analyzed (Participants) | 3 | 3 | 15 | 10 | 9
change from baseline msec
  Cycle 2 Day 1: number analyzed (Participants) | 1 | 2 | 15 | 10 | 9
  Cycle 2 Day 1 | 4.0 (NA) — Not applicable as n=1 | -14.0 (19.8) | 1.1 (23.9) | -5.1 (9.9) | 1.2 (5.3)
  Cycle 3, Day 1: number analyzed (Participants) | 3 | 2 | 12 | 5 | 7
  Cycle 3, Day 1 | 8.0 (6.0) | -12.0 (0.0) | -5.3 (26.2) | -2.8 (8.4) | -1.9 (7.5)
  Cycle 4, Day 1: number analyzed (Participants) | 1 | 2 | 8 | 1 | 7
  Cycle 4, Day 1 | 14.0 (NA) — Not applicable as n=1 | -13.0 (1.4) | -16.3 (28.4) | -10.0 (NA) — Not applicable as n=1 | -11.9 (15.7)
  Cycle 5, Day 1: number analyzed (Participants) | 1 | 2 | 5 | 2 | 5
  Cycle 5, Day 1 | -2.0 (NA) — Not applicable as n=1 | -16.0 (2.8) | -7.6 (24.5) | -11.0 (7.1) | -24.6 (7.2)
  Cycle 6, Day 1: number analyzed (Participants) | 1 | 3 | 4 | 0 | 7
  Cycle 6, Day 1 | -44.0 (NA) — Not applicable as n=1 | -19.3 (9.2) | -12.8 (21.8) |  | -3.4 (19.5)
  Cycle 7, Day 1: number analyzed (Participants) | 0 | 3 | 4 | 1 | 6
  Cycle 7, Day 1 |  | -17.3 (9.5) | -6.8 (12.0) | -2.0 (NA) — Not applicable as n=1 | -8.3 (20.9)
  Cycle 8, Day 1: number analyzed (Participants) | 1 | 0 | 3 | 1 | 5
  Cycle 8, Day 1 | 4.0 (NA) — Not applicable as n=1 |  | -5.3 (27.2) | -6.0 (NA) — Not applicable as n=1 | -9.4 (16.2)
  Cycle 9, Day 1: number analyzed (Participants) | 0 | 2 | 2 | 1 | 5
  Cycle 9, Day 1 |  | -10.0 (0.0) | -17.0 (46.7) | 6.0 (NA) — Not applicable as n=1 | 0.6 (8.5)
  Cycle 10, Day 1: number analyzed (Participants) | 1 | 1 | 3 | 0 | 2
  Cycle 10, Day 1 | -4.0 (NA) — Not applicable as n=1 | -2.0 (NA) — Not applicable as n=1 | -11.3 (30.1) |  | 1.0 (1.4)
  Cycle 11, Day 1: number analyzed (Participants) | 1 | 0 | 0 | 1 | 3
  Cycle 11, Day 1 | 4.0 (NA) — Not applicable as n=1 |  |  | 4.0 (NA) — Not applicable as n=1 | -1.7 (12.7)
  Cycle 12, Day 1: number analyzed (Participants) | 0 | 0 | 1 | 1 | 2
  Cycle 12, Day 1 |  |  | -60.0 (NA) — Not applicable as n=1 | -4.0 (NA) — Not applicable as n=1 | -5.0 (1.4)
  Cycle 13, Day 1: number analyzed (Participants) | 1 | 0 | 1 | 0 | 2
  Cycle 13, Day 1 | -2.0 (NA) — Not applicable as n=1 |  | -44.0 (NA) — Not applicable as n=1 |  | 3.0 (1.4)
  Cycle 14, Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Cycle 14, Day 1 |  |  | -54.0 (NA) — Not applicable as n=1 |  |
  Cycle 15, Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1
  Cycle 15, Day 1 | 0.0 (NA) — Not applicable as n=1 |  |  |  | -10.0 (NA) — Not applicable as n=1
  Cycle 16, Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Cycle 16, Day 1 |  |  |  |  | -2.0 (NA) — Not applicable as n=1

31. Secondary Outcome: Change From Baseline of Electrocardiogram (ECG) Endpoints: QRS Interval - Phases 1 and 2
Description: Change from baseline of ECG endpoints
  QRS interval measured in milliseconds (msec)
Time Frame: From first dose until a minimum follow-up of up to 2 months
Population: All treated participants
Measure: Mean (Standard Deviation); unit: change from baseline msec
Arm/Group | ULO 600mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph2 | ULO 1000mg + LDAC - Ph2 | LDAC - Ph2
Number analyzed (Participants) | 3 | 3 | 15 | 13 | 9
change from baseline msec
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 2 | 15 | 13 | 9
  Cycle 2 Day 1 | 0.0 (5.7) | -2.0 (5.7) | 5.1 (11.3) | 0.5 (9.6) | 4.8 (12.5)
  Cycle 3, Day 1: number analyzed (Participants) | 3 | 2 | 13 | 6 | 7
  Cycle 3, Day 1 | 3.3 (7.6) | -2.0 (5.7) | -1.3 (7.6) | 2.0 (3.4) | 1.4 (8.2)
  Cycle 4, Day 1: number analyzed (Participants) | 1 | 2 | 9 | 3 | 7
  Cycle 4, Day 1 | 0.0 (NA) — Not applicable as n=1 | 1.0 (1.4) | 2.7 (8.8) | -3.3 (6.1) | 6.4 (16.1)
  Cycle 5, Day 1: number analyzed (Participants) | 1 | 2 | 6 | 2 | 5
  Cycle 5, Day 1 | 8.0 (NA) — Not applicable as n=1 | -4.0 (2.8) | 1.8 (9.5) | 2.0 (5.7) | -1.4 (2.4)
  Cycle 6, Day 1: number analyzed (Participants) | 1 | 3 | 4 | 0 | 7
  Cycle 6, Day 1 | 6.0 (NA) — Not applicable as n=1 | -2.7 (4.2) | -1.8 (6.2) |  | 5.4 (14.7)
  Cycle 7, Day 1: number analyzed (Participants) | 0 | 3 | 4 | 1 | 6
  Cycle 7, Day 1 |  | -2.7 (4.2) | -3.3 (7.0) | -10.0 (NA) — Not applicable as n=1 | -1.5 (4.9)
  Cycle 8, Day 1: number analyzed (Participants) | 1 | 0 | 3 | 1 | 5
  Cycle 8, Day 1 | 2.0 (NA) — Not applicable as n=1 |  | 0.7 (2.3) | -8.0 (NA) — Not applicable as n=1 | 2.6 (6.9)
  Cycle 9, Day 1: number analyzed (Participants) | 0 | 2 | 2 | 1 | 5
  Cycle 9, Day 1 |  | -1.0 (1.4) | -2.0 (8.5) | -6.0 (NA) — Not applicable as n=1 | 0.0 (3.2)
  Cycle 10, Day 1: number analyzed (Participants) | 1 | 1 | 3 | 0 | 2
  Cycle 10, Day 1 | 2.0 (NA) — Not applicable as n=1 | -4.0 (NA) — Not applicable as n=1 | -2.3 (8.6) |  | 9.5 (4.9)
  Cycle 11, Day 1: number analyzed (Participants) | 1 | 0 | 0 | 1 | 3
  Cycle 11, Day 1 | 6.0 (NA) — Not applicable as n=1 |  |  | -4.0 (NA) — Not applicable as n=1 | 9.0 (7.5)
  Cycle 12, Day 1: number analyzed (Participants) | 0 | 0 | 1 | 1 | 2
  Cycle 12, Day 1 |  |  | -6.0 (NA) — Not applicable as n=1 | -8.0 (NA) — Not applicable as n=1 | 10.0 (5.7)
  Cycle 13, Day 1: number analyzed (Participants) | 1 | 0 | 1 | 0 | 2
  Cycle 13, Day 1 | 2.0 (NA) — Not applicable as n=1 |  | -12.0 (NA) — Not applicable as n=1 |  | 3.5 (10.6)
  Cycle 14, Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Cycle 14, Day 1 |  |  | -10.0 (NA) — Not applicable as n=1 |  |
  Cycle 15, Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1
  Cycle 15, Day 1 | 6.0 (NA) — Not applicable as n=1 |  |  |  | 8.0 (NA) — Not applicable as n=1
  Cycle 16, Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Cycle 16, Day 1 |  |  |  |  | 7.0 (NA) — Not applicable as n=1

32. Secondary Outcome: Change From Baseline of Electrocardiogram (ECG) Endpoints: QT Interval - Phases 1 and 2
Description: Change from baseline of ECG endpoints
  QT interval measured in milliseconds (msec)
Time Frame: From first dose until a minimum follow-up of up to 2 months
Population: All treated participants
Measure: Mean (Standard Deviation); unit: change from baseline msec
Arm/Group | ULO 600mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph2 | ULO 1000mg + LDAC - Ph2 | LDAC - Ph2
Number analyzed (Participants) | 3 | 3 | 15 | 13 | 9
change from baseline msec
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 2 | 15 | 13 | 9
  Cycle 2 Day 1 | -41.0 (94.8) | -5.0 (7.1) | 4.5 (25.5) | 10.4 (50.1) | 14.2 (33.7)
  Cycle 3, Day 1: number analyzed (Participants) | 3 | 2 | 13 | 6 | 7
  Cycle 3, Day 1 | 10.0 (36.7) | 7.0 (29.7) | -15.4 (30.6) | -10.7 (41.3) | 13.7 (41.7)
  Cycle 4, Day 1: number analyzed (Participants) | 1 | 2 | 9 | 3 | 7
  Cycle 4, Day 1 | -60.0 (NA) — Not applicable as n=1 | 35.0 (32.5) | 10.1 (22.8) | -12.7 (104.3) | -1.4 (47.9)
  Cycle 5, Day 1: number analyzed (Participants) | 1 | 2 | 6 | 2 | 5
  Cycle 5, Day 1 | 12.0 (NA) — Not applicable as n=1 | 13.0 (15.6) | 2.2 (32.1) | -5.0 (26.9) | -27.6 (75.5)
  Cycle 6, Day 1: number analyzed (Participants) | 1 | 3 | 4 | 0 | 7
  Cycle 6, Day 1 | 2.0 (NA) — Not applicable as n=1 | 6.0 (26.9) | -11.8 (19.1) |  | -3.6 (39.3)
  Cycle 7, Day 1: number analyzed (Participants) | 0 | 3 | 4 | 1 | 6
  Cycle 7, Day 1 |  | 29.3 (20.0) | 11.8 (13.6) | -8.0 (NA) — Not applicable as n=1 | -8.8 (28.3)
  Cycle 8, Day 1: number analyzed (Participants) | 1 | 0 | 3 | 1 | 5
  Cycle 8, Day 1 | 2.0 (NA) — Not applicable as n=1 |  | 2.0 (2.0) | -24.0 (NA) — Not applicable as n=1 | 0.8 (35.5)
  Cycle 9, Day 1: number analyzed (Participants) | 0 | 2 | 2 | 1 | 5
  Cycle 9, Day 1 |  | 37.0 (9.9) | -23.0 (21.2) | -14.0 (NA) — Not applicable as n=1 | -24.4 (23.0)
  Cycle 10, Day 1: number analyzed (Participants) | 1 | 1 | 3 | 0 | 2
  Cycle 10, Day 1 | 6.0 (NA) — Not applicable as n=1 | 14.0 (NA) — Not applicable as n=1 | -18.3 (18.6) |  | -6.0 (11.3)
  Cycle 11, Day 1: number analyzed (Participants) | 1 | 0 | 0 | 1 | 3
  Cycle 11, Day 1 | 16.0 (NA) — Not applicable as n=1 |  |  | -22.0 (NA) — Not applicable as n=1 | 7.0 (2.6)
  Cycle 12, Day 1: number analyzed (Participants) | 0 | 0 | 1 | 1 | 2
  Cycle 12, Day 1 |  |  | -4.0 (NA) — Not applicable as n=1 | -36.0 (NA) — Not applicable as n=1 | -6.5 (27.6)
  Cycle 13, Day 1: number analyzed (Participants) | 1 | 0 | 1 | 0 | 2
  Cycle 13, Day 1 | 20.0 (NA) — Not applicable as n=1 |  | -40.0 (NA) — Not applicable as n=1 |  | -15.0 (18.4)
  Cycle 14, Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0
  Cycle 14, Day 1 |  |  | -44.0 (NA) — Not applicable as n=1 |  |
  Cycle 15, Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1
  Cycle 15, Day 1 | 36.0 (NA) — Not applicable as n=1 |  |  |  | -19.0 (NA) — Not applicable as n=1
  Cycle 16, Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Cycle 16, Day 1 |  |  |  |  | -105.0 (NA) — Not applicable as n=1

33. Secondary Outcome: Overall Survival (OS) - Phases 1 and 2
Description: OS is defined as the time between the first date of treatment and the date of death due to any cause. A participant who has not died was be censored at the last known alive date.
Time Frame: From first dose until a minimum follow-up of up to 2 months
Population: All treated participants for phase 2. Phase 1 OS data not collected.
Measure: Median (Full Range); unit: Months
Arm/Group | ULO 600mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph1 | ULO 800mg + LDAC - Ph2 | ULO 1000mg + LDAC - Ph2 | LDAC - Ph2
Number analyzed (Participants) | 0 | 0 | 26 | 14 | 22
Months |  |  | 3.3 [1.8 to 8.7] | 3.0 [1.8 to 4.7] | 6.9 [1.6 to 12.7]

ADVERSE EVENTS:
Time Frame: Includes on-treatment events from first dose to within 100 days of last dose
Description: At the end of the randomized treatment period, 6 participants in the LDAC only arm proceeded to treatment with added ulocuplumab. All 6 of the participants who added ulocuplumab following completion of LDAC only treatment have discontinued treatment. The safety data for these 6 participants are represented in the LDAC arm below.
Groups:
- Ulo 600mg+LDAC: Ulocuplumab (ULO) at 600mg + low dose cytarabine (LDAC) - Phase 1 (Ph1)
- Ulo 800mg+LDAC: Ulocuplumab (ULO) at 800mg + low dose cytarabine (LDAC) - Phase 1 (Ph1)
- Ulocuplumab 800mg + LDAC 20mg BID: Ulocuplumab (ULO) at 800mg + low dose cytarabine (LDAC) - Phase 2 (Ph2)
- Ulocuplumab 1000mg + LDAC 20mg BID: Ulocuplumab (ULO) at 1000mg + low dose cytarabine (LDAC) - Phase 2 (Ph2)
- LDAC 20mg BID: Low dose cytarabine (LDAC) - Phase 2 (Ph2) Participants in the LDAC only arm were permitted to add ulocuplumab 800 mg into their treatment regimen if they did not achieve complete remission (CR or complete remission with incomplete blood count recovery [CRi]) confirmed by blast count reduction after 4 treatment cycles or if they relapsed after achieving complete remission.
Arm/Group | Ulo 600mg+LDAC | Ulo 800mg+LDAC | Ulocuplumab 800mg + LDAC 20mg BID | Ulocuplumab 1000mg + LDAC 20mg BID | LDAC 20mg BID
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 19/26 | 10/14 | 16/22
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 21/26 | 8/14 | 15/22
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 25/26 | 14/14 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ulo 600mg+LDAC (N=3) | Ulo 800mg+LDAC (N=3) | Ulocuplumab 800mg + LDAC 20mg BID (N=26) | Ulocuplumab 1000mg + LDAC 20mg BID (N=14) | LDAC 20mg BID (N=22)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 8 | 5 | 6
Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac disorder (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Catheter site haemorrhage (General disorders) | 0 | 0 | 1 | 0 | 0
Complication associated with device (General disorders) | 0 | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 3 | 0 | 1
Pneumonia fungal (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 3 | 2 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Amylase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Epstein-Barr virus associated lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 5 | 2 | 6
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Neurogenic shock (Vascular disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ulo 600mg+LDAC (N=3) | Ulo 800mg+LDAC (N=3) | Ulocuplumab 800mg + LDAC 20mg BID (N=26) | Ulocuplumab 1000mg + LDAC 20mg BID (N=14) | LDAC 20mg BID (N=22)
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 11 | 3 | 8
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 3 | 5 | 4 | 7
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 4 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 6 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 2 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 3
Tachycardia (Cardiac disorders) | 0 | 0 | 2 | 0 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 10 | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 6 | 3 | 5
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 2
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 6 | 8 | 6
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1
Periodontal disease (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 3 | 5 | 3 | 4
Vomiting (Gastrointestinal disorders) | 1 | 1 | 4 | 1 | 3
Asthenia (General disorders) | 0 | 0 | 3 | 0 | 2
Catheter site erythema (General disorders) | 0 | 0 | 2 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 3 | 2
Early satiety (General disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 5 | 4 | 5
Generalised oedema (General disorders) | 0 | 0 | 1 | 1 | 0
Malaise (General disorders) | 0 | 0 | 3 | 0 | 1
Mass (General disorders) | 0 | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 2 | 2 | 0
Oedema peripheral (General disorders) | 1 | 2 | 6 | 1 | 4
Pyrexia (General disorders) | 2 | 2 | 8 | 5 | 5
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hepatic congestion (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 2 | 0 | 1
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Hypersensitivity (Immune system disorders) | 1 | 1 | 1 | 2 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 1 | 3
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 1 | 2
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 2
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 2
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 2 | 1 | 2
Amylase increased (Investigations) | 0 | 0 | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 3 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 2
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 1 | 0
Lipase increased (Investigations) | 1 | 0 | 2 | 0 | 2
Neutrophil count decreased (Investigations) | 2 | 0 | 3 | 1 | 6
Platelet count decreased (Investigations) | 2 | 3 | 6 | 4 | 8
Troponin T increased (Investigations) | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 2
White blood cell count decreased (Investigations) | 0 | 0 | 5 | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 3 | 2 | 4
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 3 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 4 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 3
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0 | 2
Headache (Nervous system disorders) | 0 | 0 | 3 | 3 | 2
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 7 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Renal tubular disorder (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Genital ulceration (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 6 | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 4 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 3 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 2 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 3 | 2 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-07-27): https://cdn.clinicaltrials.gov/large-docs/63/NCT02305563/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/63/NCT02305563/SAP_001.pdf